CLINICAL TRIAL: NCT02714296
Title: Phase IV Prospective Sinle Center Randomised Three-arm Controlled Study Evaluating the Effectiveness of Colon Preparation for Endoscopy Using Specialized Clinical Nutrition
Brief Title: Evaluating the Effectiveness of Colon Preparation for Endoscopy Using Specialized Clinical Nutrition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nutricia Advanced (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nutricia-001
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Colonoscopy
Keywords: colon preparation for endoscopy; enteral feeding; sip feeding; nutridrink; nutridrink compact protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group Nutridrink 200ml (Active Comparator): 50 patients: two days before the investigation is assigned to a diet with the use of specialized clinical nutrition Nutridrink 200 ml 6 bottles per day as a sole source of nutrition. On the day of the colonoscopy, as breakfast, allowed Nutridrink 1-2 bottles
  Interventions: Drug: Nutridrink 200 ml
- Group Nutridrink compact protein (Active Comparator): two days before the study is assigned diet with the addition of specialized clinical nutrition Nutridrinc compact protein 125 ml 2 bottles per day. On the day of the colonoscopy, as breakfast, allowed Nutridrink compact protein 1-2 bottles
  Interventions: Dietary Supplement: Nutridrink compact protein
- Group control (No Intervention): only diet without receiving specialized nutrition

INTERVENTIONS:
Drug: Nutridrink 200 ml — Nutridrink 200 ml 6 bottles per day as a sole source of nutrition. On the day of the colonoscopy, as breakfast, allowed Nutridrink 1-2 bottles
  Arms: Group Nutridrink 200ml
Dietary Supplement: Nutridrink compact protein — 2 bottles per day. On the day of the colonoscopy, as breakfast, allowed Nutridrink compact protein 1-2 bottles
  Arms: Group Nutridrink compact protein

SUMMARY:
This study is an open, prospective, comparative diagnostic studies aimed at improving the colonoscopy results, by optimizing the way of preparation for endoscopy

DETAILED DESCRIPTION:
Objective: to improve the quality of bowel preparation for endoscopy.

Research objectives:

1. Compare the three methods of colon preparation for endoscopy
2. To develop a rational strategy of preparing patients for endoscopy on the basis of the data obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years with the recommendation to conduct a diagnostic colonoscopy
2. Absence of contraindications to the use of specialized clinical nutrition products

Exclusion Criteria:

1. Conditions which are contraindicated for colonoscopy:

   * The acute phase of cerebrovascular accident
   * Acute myocardial infarction
   * severe cardiovascular, pulmonary insufficiency and mixed
   * Violations of the cardiac rhythm (paroxysmal bradyarrhythmia, atrial fibrillation with atrial fibrillation or paroxysmal atrial fibrillation, severe transverse heart block)
   * Severe clinical forms (fulminant) inflammatory diseases of the colon (ulcerative colitis, Crohn's disease, ischemic colitis, radiation colitis, diverticulitis)
   * Aortic aneurysm or heart
   * Acute inflammatory infiltrates abdominal cavity (including diverticulitis)
   * Suspicion of abscess of the abdominal cavity
   * Peritonitis
   * Hepatosplenomegaly
   * Tense ascites
   * hydrothorax, hydropericardium
   * Severe blood coagulation
   * Hemorrhagic vasculitis
2. Pregnancy
3. The patient's refusal to participate in the study
4. Intolerance of specialized clinical nutrition products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
the degree of preparation in the colonoscopy (Chicago or Boston scale). | before colonoscopy

SECONDARY OUTCOMES:
tolerability | before colonoscopy
  Visual analog scale assessment of tolerability of the preparation to the study

CONTACTS AND LOCATIONS:
Overall Officials: Elena Volkova, Study Chair
Locations (1):
- ГНЦ колопроктологии, Moscow, Russia